CLINICAL TRIAL: NCT05154981
Title: Partners in School: Promoting Continuity Across Home and School for Children with Autism by Improving Parent-Teacher Communication During the Transition to School
Brief Title: Partners in School: Promoting Continuity Across Home and School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gazi Azad, Research Scientist and Assistant Professor, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8302; 5K23MH119331-04 (NIH)
Record Dates: First submitted 2021-11-17; First posted 2021-12-13 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Schools

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Partners in School with Education Communication Skills (ECS) Training (Experimental): Parents and teachers in the experimental condition will receive Partners in School with communication training.
  Interventions: Behavioral: Education communication skills (ECS) training; Behavioral: Partners in School
- Partners in School without Education Communication Skills (ECS) Training (Active Comparator): Parents and teachers in the control condition will receive Partners in School without communication training.
  Interventions: Behavioral: Partners in School

INTERVENTIONS:
Behavioral: Education communication skills (ECS) training — Education communication skills (ECS) training videos were developed from LEAPS (Listen, Educate, Assess, Partner and Support), a set of 10- to 20- sec videos that help patients and physicians communicate health concerns and treatment plans to each other. ECS training videos target parent-teacher communication during the transition to school for children with autism.
  Arms: Partners in School with Education Communication Skills (ECS) Training
Behavioral: Partners in School — Partners in School is a problem-solving consultation that encourages parents and teachers to implement the same evidence-based interventions across home and school

SUMMARY:
Partners in School is a collection of implementation strategies (e.g., communication training, problem-solving consultation) to help parents/primary caregivers and teachers of children with autism spectrum disorder implement the same practices across home and school.

DETAILED DESCRIPTION:
We recruited a total of 48 participants (N=22 parent-teacher dyads) from urban and suburban public schools in New York, New Jersey, and Connecticut. Teachers were matched on years of teaching experience (0-2 years, 3-5 years, 5-10 years, or 11+ years), and then randomized to the experimental condition or the control condition. The experimental condition had 13 parent-teacher dyads (N=26 participants) and the control condition had 11 parent-teacher dyads (N=22 participants). The experimental condition included the five steps of Partners in School including the pre-consultation phone interview, web-based communication skills training for the parent or teacher through School Talk, in-person parent-teacher conference, three weeks of implementing the same intervention with the student at home (by parents) and school (by the teacher), and a post-consultation phone interview. Parents and teachers also completed surveys at the beginning and end of Partners in School. The control condition had the same experiences but the parents/teachers in that condition did not receive communication skills training through School Talk. One of the key outcomes is that recruitment, randomization, condition protocols, retention, and assessment of Partners in School with School Talk is feasible and acceptable. These findings are significant to the scientific field because they suggest that researchers can partner with public schools and train parents and teachers to communicate and collaborate effectively in order to double the dosage, intensity, and impact of evidenced-based practices for young children on the autism spectrum disorder (ASD).

ELIGIBILITY:
Inclusion Criteria:

1. Must be parent/primary caregiver or full-time, lead teacher
2. Must have or teach preschool, pre- kindergarten, kindergarten, or 1st grade child with ASD
3. Must have or teach child with ASD that can see and hear
4. Access to internet via wifi-enabled phone, tablet, or computer
5. Must be English or Spanish speaking
6. An active email -

Exclusion Criteria:

1. Parents with younger (less than preschool) or older children (in 2nd grade or above)
2. Teachers who teach older than 1st grade.
3. Teaching assistants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Adapted LEAPS Questionnaire about ECS training (A-LEAPS) | baseline
  The A-LEAPS will be an 18-item parent questionnaire (adapted patient form) and a 23-item teacher questionnaire (adapted physician form). At the baseline self-assessment, parents and teachers will be asked to report on their communication practices using never, sometimes, or always used. At the post-consultation self-assessment, they will be asked to again reflect on their communication practices, but this time with the specific Partners in School parent-teacher consultation meeting just completed. An example item is, "I set an agenda for the meeting so that I am sure we get to all the things I want to cover."
Adapted LEAPS Questionnaire about ECS training (A-LEAPS) | at study completion, an average of 10 weeks
  The A-LEAPS will be an 18-item parent questionnaire (adapted patient form) and a 23-item teacher questionnaire (adapted physician form). At the baseline self-assessment, parents and teachers will be asked to report on their communication practices using never, sometimes, or always used. At the post-consultation self-assessment, they will be asked to again reflect on their communication practices, but this time with the specific Partners in School parent-teacher consultation meeting just completed. An example item is, "I set an agenda for the meeting so that I am sure we get to all the things I want to cover."
Parent-Teacher Relationship Scale-Second Edition (PTRS-II) | baseline
  The PTRS-II is a 24-item measure that examines the degree of connection felt between parent and teacher pairs, by examining joining (affiliation and support, dependability and availability, shared expectations and beliefs, and communication from the other) and communication to the other (sharing of emotion and sharing of information). A five-point Likert scale is used from almost never to almost always. An example item is, "I don't like the way this teacher talks to me."
Parent-Teacher Relationship Scale-Second Edition (PTRS-II) | at study completion, an average of 10 weeks
  The PTRS-II is a 24-item measure that examines the degree of connection felt between parent and teacher pairs, by examining joining (affiliation and support, dependability and availability, shared expectations and beliefs, and communication from the other) and communication to the other (sharing of emotion and sharing of information). A five-point Likert scale is used from almost never to almost always. An example item is, "I don't like the way this teacher talks to me."
Parent-Teacher Alliance Questionnaire (PTAQ) | baseline
  The PTAQ is a 20-item measure that assesses the degree to which parents believe they have a sound working relationship with the teacher (and vice versa). A five-point Likert scale is used from strongly agree to strongly disagree. An example item is, "My child's teacher treats me as a partner in the development of my child's education plan." It was adapted from the Parenting Alliance Inventory
Parent-Teacher Alliance Questionnaire (PTAQ) | at study completion, an average of 10 weeks
  The PTAQ is a 20-item measure that assesses the degree to which parents believe they have a sound working relationship with the teacher (and vice versa). A five-point Likert scale is used from strongly agree to strongly disagree. An example item is, "My child's teacher treats me as a partner in the development of my child's education plan." It was adapted from the Parenting Alliance Inventory
Participation in Problem Solving Scale (PPSS) | baseline
  The PPSS asks respondents to assess their problem solving competencies using 12-items. Items are rated on a five-point Likert scale from disagree very strongly to agree very strongly. An example item is, "I gathered specific information to measure this student's progress."
Participation in Problem Solving Scale (PPSS) | at study completion, an average of 10 weeks
  The PPSS asks respondents to assess their problem solving competencies using 12-items. Items are rated on a five-point Likert scale from disagree very strongly to agree very strongly. An example item is, "I gathered specific information to measure this student's progress."
Change from Baseline Fidelity (to Student Intervention Plan) at 3 weeks | daily for three weeks
  Daily home-school notes will list the steps in the student intervention plan generated during the consultation meeting. Parents and teachers will indicate whether each step was completed at home or at school, respectively. The number of intervention steps completed by parents (parent fidelity) and teachers (teacher fidelity) will be computed.
Change from Baseline Alignment (of Student Intervention Plan) at 3 weeks | daily for three weeks
  Daily home-school notes will list the steps in the student intervention plan generated during the consultation meeting. Parents and teachers will indicate whether each step was completed at home or at school, respectively. The number of steps in the student intervention plan completed by both parents and teachers will be used as the measure of continuity.

SECONDARY OUTCOMES:
Frequency and Severity Form (FSF) | baseline
  Using the FSF form, the consultant will ask parents and teachers to report on the top three concerns that they have for the child, as well as to rate the frequency and severity of each of those concerns. The frequency question asks, "How often does this occur with your child at school or at home?" The concern is rated on a five-point Likert scale ranging from rarely to always. The severity question asks, "How much does this impact your child's daily functioning at school or at home?" The concern is rated on a five-point Likert scale ranging from rarely to extremely. This measure was designed specifically for Partners in School.
Frequency and Severity Form (FSF) | at study completion, an average of 10 weeks
  Using the FSF form, the consultant will ask parents and teachers to report on the top three concerns that they have for the child, as well as to rate the frequency and severity of each of those concerns. The frequency question asks, "How often does this occur with your child at school or at home?" The concern is rated on a five-point Likert scale ranging from rarely to always. The severity question asks, "How much does this impact your child's daily functioning at school or at home?" The concern is rated on a five-point Likert scale ranging from rarely to extremely. This measure was designed specifically for Partners in School.
Pervasive Developmental Disorder Behavior Inventory (PDDBI) | baseline
  The PDDBI is an informant-based rating scale designed to assist in the assessment of children who have been diagnosed with autism. This measure has been developed to assess both problem behaviors as well as appropriate social, language, and learning/memory skills.
Pervasive Developmental Disorder Behavior Inventory (PDDBI) | at study completion, an average of 10 weeks
  The PDDBI is an informant-based rating scale designed to assist in the assessment of children who have been diagnosed with ASD. This measure has been developed to assess both problem behaviors as well as appropriate social, language, and learning/memory skills.
Goal Attainment Scaling (GAS) | daily for three weeks
  The home-school notes will assess the child's progress toward his/her pre-determined goal that will be formulated by parents and teachers during the consultation meeting. We will use an adapted goal attainment scaling (GAS), ranging from the situation got significantly worse (-2) to the situation got significantly better (+2).
Family-Professional Partnership Scale (FPPS) | baseline
  The FPPS is an 18-item measure designed to assess the extent of parent or teacher satisfaction with their partnership orientated practices using subscales about child-focused relationships and family-focused relationships. Items are rated on a five-point Likert scale ranging from very dissatisfied to very satisfied. An example question is, "How satisfied are you that your child's teacher values your opinions about your child's needs?"
Family-Professional Partnership Scale (FPPS) | at study completion, an average of 10 weeks
  The FPPS is an 18-item measure designed to assess the extent of parent or teacher satisfaction with their partnership orientated practices using subscales about child-focused relationships and family-focused relationships. Items are rated on a five-point Likert scale ranging from very dissatisfied to very satisfied. An example question is, "How satisfied are you that your child's teacher values your opinions about your child's needs?"
Self-Efficacy with Communication Form (SECF) | baseline
  The SECF is a five-item questionnaire designed to capture important constructs in the self-efficacy literature (e.g., competency, effectiveness, and confidence). Items are rated on a five-point Likert scale ranging from not at all to extremely. An example question is, "How confident are you at communicating with this student's parent?" Items were derived from prior studies on self-efficacy and are sensitive to changes in Partners in School.
Self-Efficacy with Communication Form (SECF) | at study completion, an average of 10 weeks
  The SECF is a five-item questionnaire designed to capture important constructs in the self-efficacy literature (e.g., competency, effectiveness, and confidence). Items are rated on a five-point Likert scale ranging from not at all to extremely. An example question is, "How confident are you at communicating with this student's parent?" Items were derived from prior studies on self-efficacy and are sensitive to changes in Partners in School.
Consultant Adherence | at study completion, an average of 10 weeks
  The Partners in School objective checklists will be used to evaluate the extent to which the consultant followed the necessary components of the Partners in School protocol. The checklist has separate objectives for the pre-consultation, consultation, and post-consultation. An example objective for the pre-consultation is, "Asked about the frequency of the concern."

CONTACTS AND LOCATIONS:
Overall Officials: Gazi Azad, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Research Foundation for Mental Hygiene at the New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No